CLINICAL TRIAL: NCT01918267
Title: U-Act-After: An Observational Study on Long-Term Efficacy of Tight Control RoActemra/Actemra (Tocilizumab) and/or Methotrexate in Patients With Early Rheumatoid Arthritis Who Have Participated in the U-Act-Early Study (ML22497)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28388
Record Dates: First submitted 2013-08-06; First posted 2013-08-07 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This non-interventional, observational, open-label multi-center follow-up study of patients from the U-Act-Early trial (ML22497) will evaluate the long-term efficacy and safety of starting tight control treatment with RoActemra/Actemra (tocilizumab) and/or methotrexate in patients early in the disease followed by treatment according to standard of care in routine clinical practice in a three year follow-up, independently of what treatment the patient will be receiving.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have participated in the U-Act-Early trial (ML22497); these are adult patients (> 20 years of age) with rheumatoid arthritis.
* Patients must be willing to give written informed consent

Exclusion Criteria:

* Patients who did not participate in the U-Act-Early trial
* Patients who are drop-outs in the U-Act-Early trial due to withdrawal of consent, are lost to follow-up or are serious protocol violators

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who participated in the U Act Early study (ML22497)
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2012-04-10 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Change in Disease Activity Score (DAS28) | from baseline to Month 36

SECONDARY OUTCOMES:
Change in disability, assessed by the Dutch consensus Health Assessment Questionnaire (HAQ) | from baseline to Month 36
Measure of progressive joint destruction (vdHSS) | from baseline of U-Act-Early to Month 24 of U-Act-After
Changes in concomitant medication (especially tapering of corticosteroids) | from baseline to Months 36
Sustained remission rates/drug-free remission rates | 36 months
Dose modifications/interruptions of RA treatment | 36 months
Safety: Incidence of adverse events, adverse events of special interest and serious adverse events | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (19):
- Netherlands (19):
  - Medisch Centrum Alkmaar, Alkmaar
  - Meander Medisch Centrum; Locatie Lichtenberg, Amersfoort
  - Gelre Ziekenhuis Apeldoorn, Lokatie Lukas; Afdeling Interne Geneeskunde, Apeldoorn
  - Amphia Ziekenhuis, Breda
  - Rivas Zorggroep, Locatie Beatrixziekenhuis; Reumatologie, Gorinchem
  - Groene Hart Ziekenhuis, Gouda
  - Universitair Medisch Centrum Groningen; Department of Rheumatology, Groningen
  - Kennemer Gasthuis; Inwendige Geneeskunde, Haarlem
  - Atrium Medisch Centrum; Nephrology, Heerlen
  - Tergooiziekenhuizen, loc. Hilversum, Hilversum
  - Spaarne Ziekenhuis; Inwendige Geneeskunde, Hoofddorp
  - Medisch Centrum Leeuwarden; Reumatology, Leeuwarden
  - Academisch Ziekenhuis Leiden; Dept of Rheumatology, Leiden
  - Ijsselmeer Ziekenhuizen; Interne Geneeskunde, Lelystad
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein
  - St. Maartenskliniek, Nijmegen
  - Antonius Ziekenhuis Sneek; Department of Rheumatology, Sneek
  - University Medical Centre Utrecht; Reumatologie en Klinische Immunologie, Utrecht
  - Maartenskliniek Woerden, Woerden